CLINICAL TRIAL: NCT07106346
Title: Encapsulation-oriented Versus Timing-oriented Strategies for the Timing of Endoscopic Ultrasound-guided Drainage in Necrotizing Pancreatitis After Acute Pancreatitis: A Multicenter Randomized Controlled Trial (WONDER-03)
Brief Title: Encapsulation-oriented vs. Timing-oriented Strategies for Necrotizing Pancreatitis
Acronym: WONDER-03
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo University (Other)
Collaborators: Tokyo Women's Medical University (Other)
Responsible Party: Principal Investigator, Yousuke Nakai, Professor, Department of Gastroenterology, Tokyo Women's Medical University, Tokyo Women's Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025002P
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Walled Off Necrosis; Pancreatitis; Acute Necrotic Collection; Necrotizing Pancreatitis; Pancreatitis, Acute Necrotizing
Keywords: Endosonography; Drainage; Walled Off Necrosis; necrotizing pancreatitis; pancreatitis
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Encapsulation-Oriented Group (Experimental): The timing of endoscopic intervention for necrotizing pancreatitis is determined based on the degree of encapsulation
  Interventions: Procedure: The timing of endoscopic intervention for necrotizing pancreatitis is determined based on the degree of encapsulation
- Timing-Oriented Group (Active Comparator): EUS-guided drainage based on the interval from the onset of acute pancreatitis
  Interventions: Procedure: EUS-guided drainage based on the interval from the onset of acute pancreatitis

INTERVENTIONS:
Procedure: The timing of endoscopic intervention for necrotizing pancreatitis is determined based on the degree of encapsulation — In the encapsulation-oriented group, participants undergo EUS-guided drainage of necrotizing pancreatitis when the degree of encapsulation reaches ≥80%, as confirmed by cross-sectional imaging (preferably contrast-enhanced CT). Imaging is repeated every 7-10 days after enrollment to assess encapsulation. Once sufficient encapsulation is observed and the patient presents with symptoms such as infection, abdominal pain, GOO or biliary obstruction, endoscopic drainage is performed. Drainage is typically performed using a lumen-apposing metal stent (LAMS) placed under EUS guidance, often accompanied by placement of an external drain. Step-up therapy, including endoscopic necrosectomy or additional drainage procedures, may be used if symptoms do not improve. If the patient improves with conservative therapy before encapsulation is achieved, drainage may be deferred. Endoscopic/percutaneous interventions should, in principle, be discussed with the expert panel beforehand.
  Arms: Encapsulation-Oriented Group
Procedure: EUS-guided drainage based on the interval from the onset of acute pancreatitis — In the timing-oriented group, participants undergo EUS-guided drainage of necrotizing pancreatitis at 4 to 5 weeks after the onset of acute pancreatitis, regardless of the degree of encapsulation. Drainage is performed only in symptomatic patients who meet predefined clinical criteria, such as signs of infection, significant pain, GOO, or biliary obstruction. Imaging is performed before the procedure. The standard approach involves placing a LAMS under EUS guidance, optionally supplemented by external drains. If symptoms do not improve, step-up interventions such as endoscopic necrosectomy, percutaneous drainage may be considered. If inflammation and symptoms improve with conservative treatment (e.g., antibiotics), EUS-guided drainage may be omitted. Conversely, even before 4-5 weeks from onset, early drainage is allowed if conservative treatment is deemed insufficient by the attending physician. In principle, intervention decisions should be discussed with the expert panel.
  Arms: Timing-Oriented Group

SUMMARY:
This multicenter, randomized controlled trial (WONDER-03 study) investigates the optimal timing for endoscopic ultrasound (EUS)-guided drainage in patients with necrotizing pancreatitis. Although current guidelines recommend delaying drainage until at least four weeks after the onset of acute pancreatitis to allow for encapsulation of necrosis, recent observational data suggest that the degree of encapsulation itself may more strongly influence treatment success and safety. In this trial, patients are randomly assigned to one of two groups: an encapsulation-oriented group, in which EUS-guided drainage is performed when imaging confirms ≥80% encapsulation of the necrotic collection with symptoms, and a timing-oriented group, in which drainage is performed at four to five weeks after disease onset, regardless of encapsulation status. The primary endpoint is clinical success within 180 days, defined as both radiologic resolution of necrosis and improvement in symptoms. Secondary endpoints include adverse event rates, recurrence of fluid collections, technical and clinical success rates, and healthcare resource use. This study aims to determine whether a strategy based on encapsulation leads to better clinical outcomes than the conventional time-based approach and may help establish a new evidence-based treatment algorithm for necrotizing pancreatitis.

DETAILED DESCRIPTION:
Necrotizing pancreatitis is a severe and potentially life-threatening condition characterized by pancreatic and/or peripancreatic tissue necrosis. Endoscopic ultrasound (EUS)-guided transmural drainage has become widely adopted as a minimally invasive approach for the management of symptomatic necrotizing pancreatitis, particularly in cases of infected collections or organ compression. Traditionally, clinical guidelines have recommended delaying such drainage procedures until four weeks after the onset of acute pancreatitis, under the assumption that encapsulation of the necrotic tissue during this time enhances safety and technical success. However, this timing-based strategy lacks robust prospective validation and may not be optimal for all patients.

Recent data from multicenter cohort studies conducted in Japan have indicated that the degree of encapsulation at the time of drainage may be a more critical factor than the elapsed time since disease onset. In these studies, patients with ≥80% encapsulation demonstrated significantly higher rates of clinical success and lower complication rates compared to those with partial or no encapsulation, regardless of the timing of intervention. This observation suggests that the current standard approach, which relies solely on time from onset, may not adequately capture individual patient readiness for intervention.

The WONDER-03 study is designed as a multicenter, open-label, randomized controlled trial to compare two treatment strategies in patients with necrotizing pancreatitis. Participants are randomly assigned to either the encapsulation-oriented group or the timing-oriented group. In the encapsulation-oriented group, EUS-guided drainage is performed once imaging, preferably contrast-enhanced CT, confirms that the necrotic collection is at least 80% encapsulated and the patient presents with symptoms such as infection, abdominal pain, gastrointestinal obstruction, or biliary obstruction. In the timing-oriented group, drainage is scheduled for four to five weeks after the onset of acute pancreatitis if the patient is symptomatic, irrespective of the encapsulation status.

Eligible patients must be 18 years or older, have a diagnosis of necrotizing pancreatitis based on imaging, and be enrolled within 28 days of disease onset. Exclusion criteria include unclear onset timing, prior drainage procedures, a diagnosis of chronic pancreatitis, contraindications to endoscopic treatment, or pregnancy. Randomization is stratified by participating institution and the presence of organ failure.

The primary outcome of the study is clinical success within 180 days of randomization, defined as both a reduction in the maximum diameter of the necrotic collection to ≤2 cm on CT or MRI, and resolution of the symptoms that necessitated intervention. These may include normalization of inflammatory markers in infected cases, relief of abdominal pain or gastrointestinal obstruction, or resolution of biliary obstruction.

Secondary outcomes include the incidence of procedure-related complications, technical success of EUS drainage, time to clinical success, recurrence of pancreatic fluid collections, mortality, total number and duration of interventions, need for surgery, length of hospitalization and ICU stay, duration of antibiotic therapy, and related medical costs. In addition, long-term outcomes such as the development of diabetes, exocrine pancreatic insufficiency, sarcopenia, and pancreatic cancer will be monitored over a follow-up period of five years.

The trial also incorporates centralized oversight through an expert panel, which assists in evaluating imaging findings to confirm eligibility and encapsulation status. All procedures are performed by experienced endoscopists, and treatment protocols, including use of lumen-apposing metal stents (LAMS), necrosectomy, and step-up interventions, are standardized across sites.

By directly comparing the two strategies in a prospective, randomized setting, this study aims to generate high-quality evidence to guide clinical decision-making in the management of necrotizing pancreatitis. If encapsulation-oriented timing proves superior, it could shift clinical practice toward a more individualized, pathology-driven approach, improving patient outcomes while reducing the risk of complications and unnecessary delays in treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with necrotizing pancreatitis according to the revised Atlanta classification, confirmed by contrast-enhanced CT (plain CT or MRI may be substituted if contrast-enhanced CT is not feasible).
* Within 28 days of onset of acute pancreatitis.
* Age ≥ 18 years at the time of consent, regardless of sex.
* Provided written informed consent from the patient or a legally authorized representative after sufficient explanation.
* Patients who are either hospitalized or being followed as outpatients at participating study institutions.

Exclusion Criteria:

* Unknown date of onset of acute pancreatitis.
* Patients who have already undergone transluminal drainage with stent placement for necrotizing pancreatitis.
* Diagnosis of chronic pancreatitis.
* Patients for whom endoscopic treatment is deemed unsafe.
* Pregnant women.
* Patients deemed inappropriate for the study by the principal investigator or sub-investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate within 180 days after randomization | Six months
  Defined as reduction of necrotic collection to ≤2 cm on imaging and resolution of symptoms that required intervention (infection: at least two out of the following inflammatory indicators: body temperature, white blood cell count, and C-reactive protein, pain, GI obstruction, or jaundice).

SECONDARY OUTCOMES:
Rate of procedure-related adverse events | 5 years
  Adverse events will be classified according to the ASGE lexicon and AGREE classification.
All-cause mortality | 5 years
  Includes any death occurring during the study period.
Time to clinical success | 180 days
  Defined as the number of days between randomization and the achievement of both imaging and symptom resolution criteria.
Technical success of initial EUS-guided drainage | At the time of first EUS-guided drainage procedure
  Defined as successful drainage of necrotizing pancreatitis
Incidence of biliary or gastrointestinal stricture | 5 years
  New diagnosis of bile duct or gastrointestinal tract stricture confirmed by imaging or endoscopy.
Number of total interventions related to necrotizing pancreatitis | 5 years
  Includes all endoscopic, percutaneous, and surgical interventions performed.
Total duration of intervention procedures | 5 years
  Sum of procedural times for all interventions.
Duration of stent placement for drainage | 5 years
  Number of days a drainage stent remains in situ.
Need for surgical intervention related to necrotizing pancreatitis | 5 years
  Whether surgical drainage or necrosectomy is required, including procedural details.
Total duration of hospitalization for necrotizing pancreatitis | 5 years
  Cumulative inpatient days related to pancreatitis treatment.
Total ICU stay duration | 5 years
  Total days spent in the intensive care unit.
Total number of days of antibiotic use | 5 years
  Includes both oral and intravenous antibiotic administration.
Total cost of interventions and hospitalization | 5 years
  Calculated from procedural costs and hospitalization records.
Recurrence rate of pancreatic fluid collections (PFCs) | 5 years
  Defined as symptomatic recurrence of PFCs requiring treatment.
Time to recurrence of PFCs | 5 years
  Days between clinical success and recurrence requiring intervention.
Duration of treatment for recurrent PFCs | 5 years
  Number of days required for treatment of recurrent fluid collections.
New-onset diabetes mellitus | 5 years
  Defined by clinical diagnosis and laboratory evidence (e.g., elevated HbA1c).
Development of exocrine pancreatic insufficiency | 5 years
  Based on clinical symptoms such as steatorrhea or need for enzyme supplementation.
Initiation of pancreatic enzyme replacement therapy | 5 years
  Whether enzyme therapy is started and when.
Development of pancreatic cancer | 5 years
  Confirmed by imaging and pathology.
Development of sarcopenia | 5 years
  Based on imaging analysis of muscle mass and clinical frailty indicators.
Changes in pancreatic morphology (volume) | 5 years
  Evaluated using 3D CT analysis to measure pancreatic volume

CONTACTS AND LOCATIONS:
Overall Officials: Yousuke Nakai, Principal Investigator — Department of Gastroenterology, Tokyo Women's Medical University
Locations (36):
- Japan (36):
  - Department of Gastroenterology, Aichi Medical University, Aichi, Japan
  - Department of Gastroenterology, Graduate School of Medicine, Chiba University, Chiba, Japan
  - Department of Medicine and Bioregulatory Science, Graduate School of Medical Sciences, Kyushu University, Fukuoka, Japan
  - Department of Gastroenterology, Gifu Municipal Hospital, Gifu, Japan
  - Department of Gastroenterology, Gifu Prefectural General Medical Center, Gifu, Japan
  - First Department of Internal Medicine, Gifu University Hospital, Gifu, Japan
  - Department of Gastroenterology and Hepatology, Hokkaido University Hospital, Hokkaido, Japan
  - Division of Hepatobiliary and Pancreatic Diseases, Department of Gastroenterology, Hyogo MedicalUniversity, Hyōgo, Japan
  - Department of Gastroenterology and Neurology, Faculty of Medicine, Kagawa University, Kagawa, Japan
  - Digestive and Lifestyle Diseases, Kagoshima University Graduate School of Medical and Dental Sciences, Kagoshima, Japan
  - Department of Gastroenterology, Kameda Medical Center, Kamogawa, Japan
  - Department of Gastroenterology, St. Marianna University School of Medicine, Kanagawa, Japan
  - Department of Gastroenterology and Hepatology, Saitama Medical Center, Saitama Medical University, Kawagoe, Japan
  - Department of Gastroenterology, Teikyo University Mizonokuchi Hospital, Kawasaki, Japan
  - Division of Gastroenterology, Department of Internal Medicine, Kobe University Graduate School ofMedicine, Kobe, Japan
  - Department of Gastroenterology and Hepatology, Mie University Hospital, Mie, Japan
  - Department of Gastroenterology and Hepatology, Okayama University Hospital, Okayama, Japan
  - 2nd Department of Internal Medicine, Osaka Medical and Pharmaceutical University, Osaka, Japan
  - Department of Gastroenterology and Hepatology, Kansai Medical University Medical Center, Osaka, Japan
  - Department of Gastroenterology and Hepatology, Kindai University Faculty of Medicine, Osaka, Japan
  - Department of Gastroenterology, Shiga University of Medical Science, Shiga, Japan
  - Department of Gastroenterology, Tokyo Women's Medical University, Tokyo, Japan
  - Division of Gastroenterology and Hepatology, Department of Medicine, Nihon University School of Medicine, Tokyo, Japan
  - Department of Gastroenterology, Wakayama Medical University School of Medicine, Wakayama, Japan
  - Department of Gastroenterology and Metabolism, Nagoya City University Graduate School of Medical Sciences, Aichi, Tokyo
  - Department of Gastroenterology, Nagoya University, Aichi, Tokyo
  - Department of Gastroenterology, The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - Department of Gastroenterology, Graduate School of Medicine, Juntendo University, Bunkyō-Ku, Tokyo
  - Department of Gastroenterology, Fukuoka University, Fukuoka, Tokyo
  - Department of Gastroenterology, Kurume University, Fukuoka, Tokyo
  - Department of Gastroenterology, Matsunami General Hospital, Gifu, Tokyo
  - Department of Gastroenterology, Hiroshima University, Hiroshima, Tokyo
  - Department of Gastroenterology, JA Onomichi General Hospital, Hiroshima, Tokyo
  - Gastroenterology Center, Yokohama City University Medical Center, Kanagawa, Tokyo
  - Department of Gastrointestinal, Hepatobiliary and Pancreatic Diseases, Sendai City Medical Center (Sendai Open Hospital), Miyagi, Tokyo
  - Third Department of Internal Medicine, University of Toyama, Toyama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216